CLINICAL TRIAL: NCT00915720
Title: Implanted Loop Recorder Surveillance of Recurrent Atrial Fibrillation After Atrial Fibrillation Ablation
Brief Title: Implanted Loop Recorder Post Atrial Fibrillation Ablation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Thoracic & Cardiovascular Healthcare Foundation (Other)
Collaborators: Medtronic (Industry); AtriCure, Inc. (Industry)
Responsible Party: John H. Ip, MD FACC, Thoracic & Cardiovascular Healthcare Foundation
Other Study IDs: ILR 1208
Record Dates: First submitted 2009-06-04; First posted 2009-06-08 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Surgical Ablation; Implanted loop recorder; Atrial Fibrillation Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a pilot study to determine if implanted loop recorders can more effectively monitor atrial fibrillation recurrence after atrial fibrillation ablation.

DETAILED DESCRIPTION:
Atrial Fibrillation (AF)is the most common arrhythmia and causes significant morbidity and mortality. Treatment for AF consists of medical therapy and ablation therapy. Medical therapies can help approximately 50% of patients, the rest must resort to ablation procedures.

Ablation procedures aim to isolate the pulmonary vein from the atrial tissue electrically and can be performed either endocardially through catheters inserted through the femoral veins or epicardially through a minimal lateral thoracotomy. Both procedures are accepted as standard of care.

Recurrent AF after ablation therapy can be common and occurs in 50% of patients and could be in a form of short periods of AF or persistent AF with less or minimal symptoms. This is of significant clinical relevance as most of these AF episodes are not recognized and can lead to thromboembolic events such as stroke. However, techniques of surveillance of AF post ablation have been suboptimal. Physicians could use holter monitoring but this is limited to a short period of 24 - 48 hours. Event recorders which are external can be used but patients need to experience symptoms associated with the AF episodes in order to record the episodes.

Better AF monitoring techniques especially after AF ablation are necessary so that recognition of AF recurrence in these patient could be possible and timely anticoagulation therapy initiated may prevent strokes.

This pilot study involves implanting a loop recorder just under the skin to record cardiac rhythms 24 hours per day without any interaction by the patient. These devices are currently approved by the FDA for monitoring of syncope and will be implanted during the patients AF ablation surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgical atrial fibrillation ablation
* Patients must be 18 years or older

Exclusion Criteria:

* Patients unwilling to comply with the follow up schedule
* Pregnant or breastfeeding patients
* Patients currently participating in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgical atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-08; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Incidence/Duration of atrial and tachyarrhythmias post AF ablation | 14 months

CONTACTS AND LOCATIONS:
Overall Officials: John H Ip, MD, Principal Investigator — Thoracic & Cardiovascular Healthcare Foundation
Locations (1):
- Thoracic & Cardiovascular Healthcare Foundation, Lansing, Michigan, United States